CLINICAL TRIAL: NCT06818656
Title: The Unhide™ Project: Economic Impact Study of IVIG Treatment for PANS
Status: Completed | Type: Observational
Sponsor: Brain Inflammation Collaborative (Other)
Collaborators: Stanford University (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: BIC-2025-01
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: PANDAS; PANS; PANS Pediatric Acute-Onset Neuropsychiatric Syndrome; Pediatric Acute-onset Neuropsychiatric Syndrome (PANS); Pediatric Acute-Onset Neuropsychiatric Syndrome; Pediatric Autoimmune Neuropsychiatric Disorders Associated With Streptococcal Infections
Keywords: Natural History Study; PANDAS; PANS; IVIG; Immunomodulatory Treatments; Quality of Life; Economic Impacts; Functional Impacts; Healthcare Resource Utilization; Neuroinflammatory Disease; Patient-Reported Outcomes; Decentralized Study; Observational
MeSH Terms: conditions — Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal infections; Pediatric acute-onset neuropsychiatric syndrome; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Economic Impact Study of IVIG treatment for PANS is a part of the Unhide™ Project, which is a research initiative developed by the Brain Inflammation Collaborative. Specifically, the Unhide™ project is a collection of investigations with the overall goal of better understanding the problems with thinking and mood that can sometimes be symptoms of conditions like autoimmune disease, infection-associated chronic conditions like Long COVID, ME/CFS, PANDAS, PANS, and other illnesses. Your contribution to this research will allow us to better describe these symptoms and understand what causes them, how they develop, and how they can best be treated and prevented.

This study seeks to assess how PANDAS/PANS affects the financial well-being of families who pursue IVIG treatment, as well as the overall health and quality of life of children with the condition. By gathering data through this survey, we aim to gain important insights into the economic consequences of treating - or not treating - PANS with IVIG, including how it impacts parents' ability to work and children's ability to attend school.

Key Eligibility Criteria

* Aged 2-89, U.S. resident, fluent in English, and have access to computer and/or smartphone
* Suspected or confirmed diagnosis of PANS/PANDAS
* Have received IVIG OR have sought and/or been prescribed IVIG but have not received it

ELIGIBILITY:
Inclusion Criteria:

* Individuals who who have, or have had, a healthcare provider-diagnosed or suspected diagnosis of PANDAS and/or PANS
* Have received IVIG OR have sought and/or been prescribed IVIG but have not received it
* Fluent in English, sufficient to communicate status via the ePRO instrument as required by the protocol
* Is a U.S. resident
* Access to a computer and/or smartphone and the internet, and possessing the ability to operate those devices without assistance from another person (except that children can be assisted by their parents/guardians).

Exclusion Criteria:

* Ward of state
* Failure to meet inclusion criteria

Ages: 2 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals will be recruited through social media and various online channels.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Economic and Quality of Life Impact of IVIG treatment | Baseline
  This survey asks respondents (and/or their parent/legal guardian) about aspects of IVIG treatment related to medical encounters, treatment access, financial impacts, insurance coverage, and the functional and emotional effects of PANS/PANDAS.

CONTACTS AND LOCATIONS:
Locations (1):
- Brain Inflammation Collaborative, Delafield, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Brain Inflammation Collaborative (BIC) Research Collaborators selected by BIC will have access to data reports from registry participants, in keeping with criteria of the specific collaborative investigation.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available to BIC Research Collaborators as long as the study remains active, and for 7 years thereafter upon request.
Access Criteria: BIC Research Collaborators will be selected based on mutual interest and on BIC's assessment that the Collaborator possesses knowledge, experience, ethics, and training that will benefit interpretation of registry data, and proposes a meritorious and feasible research project in line with BIC's Research Roadmap.